CLINICAL TRIAL: NCT05171517
Title: Study on Microflora Characteristics of Pancreatic Solid Lesions Via Endoscopic Ultrasound-guided Fine Needle Aspiration/Biopsy
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, SHENGYU ZHANG, Principal Investigator, Peking Union Medical College Hospital
Other Study IDs: ZS-3264
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Carcinoma; Pancreatic Neuroendocrine Tumor; Autoimmune Pancreatitis; Microflora
Keywords: pancreatic solid lesion; microflora; fine needle aspiration/biopsy
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoma, Islet Cell; Autoimmune Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The remaining fresh tissue after sufficient specimen collected for the diagnosis acquired via EUS-FNA/B will be stored in - 80℃ fridge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study objective: To describe the microflora characteristics of the pancreatic solid lesions via the tissue acquired via the endoscopic ultrasound-guided fine needle aspiration/biopsy (EUS-FNA/B).

Study design: This is a prospective observational study.

DETAILED DESCRIPTION:
This is a prospective observational study. Patients who need EUS-FNA/B for diagnosis of pancreatic solid lesions (pancreatic cancer, chronic pancreatitis, and autoimmune pancreatitis, etc)will be successively included in this study. The EUS-FNA/B procedures will be accomplished in the standard way after the puncture site is washed with 20ml sterile saline for three times. The remaining fresh tissue after sufficient specimen collected for the diagnosis will be stored in - 80℃ fridge. DNA is extracted from all samples using the suitable kit and V4 16S rRNA gene sequencing is performed on all samples. The investigators ran "Decontam" (Davis NM, et al. Microbiome 2018;6:226) in order to identify and remove contaminant DNA sequences from the dataset. And the microbiome is analyzed with the standard methodology. The investigators tend to describe the microflora characteristics of pancreatic solid lesions and try to compare the differences between cancer and benign diseases.

This study will carry out in two stages: the preliminary stage, 10 patients will be included. If the technic success rate (successful extraction of DNA and sequencing of 16s rRNA after bioinformatical removal of potential DNA contaminations via the use of 'Decontam') is high than 50%, the successive inclusion progress [the main stage] will last for one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need EUS-FNA/B for diagnosis of pancreatic solid lesions.
* Age ≥ 18 years and < 80 years.

Exclusion Criteria:

* Including but not limited to: poor general conditions, severe cardiopulmonary disease, difficult to tolerate EUS examination; coagulation dysfunction; platelets <50×10^9/L

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who need EUS-FNA/B for diagnosis of pancreatic solid lesions.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Microflora analysis accomplished | within one month after EUS-FNA/B procedure
  successful extraction of DNA and sequencing of 16s rRNA after bioinformatical removal of potential DNA contaminations via the use of 'Decontam', and microflora result is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Aiming Yang, M.D., Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No